CLINICAL TRIAL: NCT03123770
Title: The Efficacy and Safety of Neoadjuvant Pegylated Liposomal Doxorubicin Plus Cyclophosphamide Followed by Docetaxel in Breast Cancer Patients: A Multicentric, Open-label, Non-randomized Concurrent Control, Non-inferiority Trial
Brief Title: Efficacy and Safety of Neoadjuvant DC-T in Breast Cancer Patients
Acronym: ESNDBCP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); First Affiliated Hospital of Zhejiang University (Other); Sir Run Run Shaw Hospital (Other); Women's Hospital School Of Medicine Zhejiang University (Other); Zhejiang Cancer Hospital (Other); Zhejiang Provincial People's Hospital (Other); Zhejiang Provincial Hospital of TCM (Other); First People's Hospital of Hangzhou (Other); Hangzhou Hospital of Traditional Chinese Medicine (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Ningbo No. 1 Hospital (Other); Jinhua Central Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Zhang, Dr, Zhejiang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESNDBCP
Record Dates: First submitted 2017-04-14; First posted 2017-04-21 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Neoadjuvant Chemotherapy; Pegylated liposomal doxorubicin; PLD
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; 1-dodecylpyridoxal; Cyclophosphamide; Epirubicin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DC Follow T (Experimental): Participants receive pegylated liposomal doxorubicin plus cyclophosphamide followed by docetaxel before surgery.
  Interventions: Drug: Pegylated liposomal doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- EC Follow T (Active Comparator): Participants receive epirubicin plus cyclophosphamide followed by docetaxel before surgery.
  Interventions: Drug: Cyclophosphamide; Drug: Epirubicin; Drug: Docetaxel

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin — a new kind of doxorubicin
  Other Names: PLD
  Arms: DC Follow T
Drug: Cyclophosphamide — traditional chemotherapy drug
  Other Names: C
Drug: Epirubicin — traditional chemotherapy drug used in breast cancer
  Other Names: E
  Arms: EC Follow T
Drug: Docetaxel — traditional chemotherapy drug used in breast cancer
  Other Names: T

SUMMARY:
This is a multicentric, open-label,non-randomized concurrent control, 1:1 match,non-inferiority trial that assesses the efficacy and safety of neoadjuvant chemotherapy regimen DC-T and EC-T in breast cancer patients.

DETAILED DESCRIPTION:
OBJECTIVES: Determine the efficacy and safety of neoadjuvant chemotherapy regimen DC-T and EC-T in suitable breast cancer patients.

Participants are randomized to 1 of 2 treatment arms.

1. Arm I: Participants receive pegylated liposomal doxorubicin plus cyclophosphamide followed by docetaxel before surgery.
2. Arm II: Participants receive epirubicin plus cyclophosphamide followed by docetaxel before surgery.

Patients in arms I and II will undergo physical examination, MRI, estimating of side effects every 4 cycles referring to RECIST (Response Evaluation Criteria In Solid Tumor) guideline. To adjust for potential bias, patients in DC-T arm were matched 1:1 to patients in the EC-T arm based on Her-2 and ER status. After finishing 8 cycles of neoadjuvant chemotherapy, every patient will receive mastectomy or breast-conserving surgery and then assess the pCR rate of primary lesion and axillary lymph nodes. Adjuvant radiotherapy and endocrine therapy will be taken if necessary. Every patient will be followed-up for five years to monitor survival condition.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged : 18~70 years.
2. WHO (ECOG) performance status 0-2.
3. Patients who have read and understand the informed consent form and have given written informed consent.
4. Diagnosed as invasive breast cancer by core biopsy
5. Diagnosed pre-surgically as (cTNM Staging)Stage II-III and suit for neoadjuvant chemotherapy.
6. Patients had previously not received chemotherapy，radiotherapy or biotherapy.
7. Normal organ function，meeting the requirement of laboratory testing below:

   * WBC≥4.0×109/L,
   * NEU≥1.5×109/L,
   * PLT≥100×109/L,
   * HB ≥10g/dL,
   * Scr≤1.5× ULN,
   * AST ≤2.5×ULN,
   * ALT ≤2.5×ULN,
   * TDIL≤1.5×ULN.
8. Patients with measurable lesion assessed by imaging using the RECIST (Response Evaluation Criteria In Solid Tumor) guideline，（long diameter of primary lesion ≥1cm or minor diameter of lymph node ≥1.5cm）；

Exclusion Criteria:

1. Pregnant or lactating women were excluded.
2. History of receiving organ transplantation（including Autologous bone marrow transplantation and peripheral hematopoietic stem-cell transplantation).
3. Dysfunction of peripheral nerve system caused by other diseases or history of either severe mental disorder or central nervous system disorders.
4. Uncontrolled infection or severe peptic ulcer need treatment.
5. Severe hepatic disease（such as hepatic cirrhosis),nephrosis,respiratory disease or uncontrolled diabetes.
6. Patients with malignancies (other than breast cancer) within the last 5 years, except for adequately treated in situ carcinoma of the cervix or basal cell carcinoma of the skin.
7. Significant abnormal EKG or cardiac disease with drastic symptoms like congestive heart failure or severe coronary disease or uncontrolled arrhythmia or myocardial infarction within 12 months or NYHA level III-IV or LVEF<55% .
8. Be allergic to test drugs.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | 5 years
  The pathological complete response rate of primary lesion and axillary lymph nodes

SECONDARY OUTCOMES:
Side effects | 5 years
  Determine side effects of these drugs like cardiotoxicity ,hematological toxicity，gastrointestinal symptoms and so on.
Overall survival | 5 years
  Determine the overall survival at 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Huang Jian, Dr, Study Chair — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- Cancer institute, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] O'Brien ME, Wigler N, Inbar M, Rosso R, Grischke E, Santoro A, Catane R, Kieback DG, Tomczak P, Ackland SP, Orlandi F, Mellars L, Alland L, Tendler C; CAELYX Breast Cancer Study Group. Reduced cardiotoxicity and comparable efficacy in a phase III trial of pegylated liposomal doxorubicin HCl (CAELYX/Doxil) versus conventional doxorubicin for first-line treatment of metastatic breast cancer. Ann Oncol. 2004 Mar;15(3):440-9. doi: 10.1093/annonc/mdh097. PMID 14998846
- [Background] Vici P, Pizzuti L, Gamucci T, Sergi D, Conti F, Zampa G, Del Medico P, De Vita R, Pozzi M, Botti C, Di Filippo S, Tomao F, Sperduti I, Di Lauro L. Non-pegylated liposomal Doxorubicin-cyclophosphamide in sequential regimens with taxanes as neoadjuvant chemotherapy in breast cancer patients. J Cancer. 2014 Apr 25;5(6):398-405. doi: 10.7150/jca.9132. eCollection 2014. PMID 24847380
- [Background] Gil-Gil MJ, Bellet M, Morales S, Ojeda B, Manso L, Mesia C, Garcia-Martinez E, Martinez-Janez N, Mele M, Llombart A, Pernas S, Villagrasa P, Blasco C, Baselga J. Pegylated liposomal doxorubicin plus cyclophosphamide followed by paclitaxel as primary chemotherapy in elderly or cardiotoxicity-prone patients with high-risk breast cancer: results of the phase II CAPRICE study. Breast Cancer Res Treat. 2015 Jun;151(3):597-606. doi: 10.1007/s10549-015-3415-2. Epub 2015 May 16. PMID 25981896
- [Background] Uriarte-Pinto M, Escolano-Pueyo A, Gimeno-Ballester V, Pascual-Martinez O, Abad-Sazatornil MR, Agustin-Ferrandez MJ. Trastuzumab, non-pegylated liposomal-encapsulated doxorubicin and paclitaxel in the neoadjuvant setting of HER-2 positive breast cancer. Int J Clin Pharm. 2016 Apr;38(2):446-53. doi: 10.1007/s11096-016-0278-5. Epub 2016 Mar 7. PMID 26951122